CLINICAL TRIAL: NCT05126901
Title: Randomised, Open-label, Active-controlled, Multicentre, Comparative Study to Evaluate the Safety and Efficacy of Ferric Maltol (Iron (III)-Maltol Complex) (ST10) Oral Suspension Compared to Ferrous Sulfate Oral Liquid in Children and Adolescents Aged 2 to 17 Years With Iron-deficiency Anaemia, Incorporating a Single Arm Study in Infants Aged 1 Month to Less Than 2 Years
Brief Title: Evaluate the Safety and Efficacy of Ferric Maltol Oral Suspension vs. Ferrous Sulfate Oral Liquid in Children and Adolescents Aged 2 to 17 Years With Iron-deficiency Anaemia, With a Single Arm Study in Infants Aged 1 Month to Less Than 2 Years
Acronym: FORTIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shield Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST10-01-305
Record Dates: First submitted 2021-10-27; First posted 2021-11-19 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Anemia; Iron-deficiency
Keywords: Anemia; Iron-Deficiency
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — ferric maltol; ferric trimaltol; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: The study will include 98 subjects in the 2 - 17 years age group, randomised 1:1 between ferric maltol and ferrous sulfate: 49 in each treatment group. The study will also include up to 12 subjects in the 1 month to less than 2 years age group. If less than 91 subjects in total have been randomized when 32 ferric maltol subjects have completed, then an interim analysis will be conducted. If significant, the study will stop recruitment. If not significant, the study will continue until 54 subjects have been recruited in the ferric maltol arm.
Masking Description: 12 weeks open label treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 month to 2 year old subjects (infants) (Experimental): Subjects aged 1 month to less than 2 years will enter a Pre-assignment phase: baseline urine samples are collected and subjects will take a single dose of 0.1 ml/kg ferric maltol suspension. Further 3 samples up to 12h will be taken.
  Subjects showing evidence of absorption, metabolism and elimination of maltol will enter the treatment phase and be assigned to the ferric maltol arm.
  The first 6 subjects screened will perform the pre-assignment PK phase. After review by the investigator, and medical monitors , if Maltol Glucuronide is shown to be adequately eliminated, timepoint 20-24 hrs (+ 4hrs) will not be performed on subsequent subjects.
  Subjects will be assigned to receive ferric maltol oral suspension and start the 0.1 ml/kg BID dose on V2 and continue for 7-10 days. On V3 they will perform the same PK assessments as on Pre-assignment PK visit.
  Interventions: Drug: Ferric Maltol
- 2 to 17 year old subjects - Ferric Maltol (Experimental): Subjects aged 2-17 will be randomised 1:1 to receive ferric maltol oral suspension or ferrous sulfate oral liquid.
  The first 12 subjects randomised to ferric maltol in each age sub-group (2 - 9 yrs, 10 - 17 yrs respectively) will enter a PK phase with 2 PK days.
  Following PK Day 2 subjects will continue until Week 12. Once the 18 subjects in each age subgroup have finished their PK visits, they will continue until week 12.
  Ferrous sulfate 125 mg/ml (25 mg elemental iron) or equivalent dose will be used for all children/adolescents. To maximise the iron replenishment for subjects within this group as well; aged 2 - 17 yrs will be dosed 6 mg/kg to the maximum of 4 ml BID.
  Subjects randomised to ferrous sulfate oral liquid will not need to complete the PK period.
  Interventions: Drug: Ferric Maltol
- 2 to 17 year old subjects - Ferrous Sulfate (Active Comparator): Subjects aged 2-17 will be randomised 1:1 to receive ferric maltol oral suspension or ferrous sulfate oral liquid.
  Ferrous sulfate 125 mg/ml (25 mg elemental iron) or equivalent dose will be used for all children/adolescents. To maximise the iron replenishment for subjects within this group as well; aged 2 - 17 yrs will be dosed 6 mg/kg to the maximum of 4 ml BID.
  Subjects randomised to ferrous sulfate oral liquid will not need to complete the PK period.
  Interventions: Drug: Ferrous sulfate

INTERVENTIONS:
Drug: Ferric Maltol — Ferric maltol oral suspension: 150 ml amber glass bottle with graduated syringe and adaptor. Oral suspension containing 30 mg elemental iron, in the form of 231.5 mg ferric maltol, in 5 ml suspension
  Study dosage: The dose of ferric maltol oral suspension that will be administered for children aged 1 month to < 2 yrs: 0.1 ml/kg BID, 2 to - 11 yrs: 2.5 ml BID, 12-17 yrs: 5 ml BID.
  Other Names: Feraccru; Ferric Trimaltol; ST10; ST10-01
  Arms: 1 month to 2 year old subjects (infants); 2 to 17 year old subjects - Ferric Maltol
Drug: Ferrous sulfate — Ferrous sulfate 125 mg/ml (25 mg/ml elemental iron) oral liquid : 15 ml glass bottle.
  Study dosage: For ferrous sulfate oral liquid, the dose administered will be for children and adolescents aged 2 years to 17 yrs: 6 mg/kg to the maximum of 4 ml BID.
  Arms: 2 to 17 year old subjects - Ferrous Sulfate

SUMMARY:
The objective of the study is to compare the safety and gastrointestinal tolerability of ferric maltol oral suspension and ferrous sulfate oral liquid in children and adolescents aged 2 years to 17 years, and assess the safety and tolerability of ferric maltol oral suspension in children 1 month to less than 2 years, in the treatment of iron deficiency anaemia during the 12 weeks treatment period.

DETAILED DESCRIPTION:
The study is a randomised, Open-label, Active-controlled, Multicentre, Comparative Study to Evaluate the Safety and Efficacy of Ferric Maltol (Iron (III)-Maltol Complex) (ST10) Oral Suspension Compared to Ferrous Sulfate Oral Liquid in Children and Adolescents Aged 2 to 17 Years With Iron-deficiency Anaemia, Incorporating a Single Arm Study in Infants Aged 1 Month to Less Than 2 Years.

Approximately 110 male and female children from 1 month to 17 years of age, with iron deficiency anaemia. If less than 91 subjects in total have been randomized when 32 ferric maltol subjects have completed, then an interim analysis will be conducted.

Subjects aged 2 to 17 years will be 1:1 randomised to ferric maltol and ferrous sulfate, with 49 subjects in each arm. Subjects then will be further divided into 2 age groups: 2 yrs - 9 yrs and 10 yrs -17 yrs. A minimum of 18 subjects must be recruited into the 2 yrs - 9 yrs and 10 yrs - 17 yrs age groups and a minimum of 25% of either sex must be recruited.

A maximum of 12 subjects will be recruited in the 1 month to less than 2 years age group. They will only be assigned to the ferric maltol group, once there is evidence of absorption, of serum iron and elimination of maltol from the Pre-assignment PK samples by showing urine maltol return to baseline, or to a low level, confirming no accumulation of maltol or maltol glucuronide, they will continue on to the 12 weeks treatment phase.

Design: The study will comprise of the following stages:

* Screening: within 14 days prior to randomisation for each subject
* Pre-assignment PK phase: only applicable for subjects aged 1 month to less than 2 years. Up to 21 days from Screening.
* Randomised treatment: 12 weeks open label treatment
* Assigned treatment phase 12 weeks open label treatment for ferric maltol children aged 1 month to less than 2 years
* End of study: Week 12 visit
* Post-treatment safety follow-up: 10-14 days following study completion of the treatment period or premature discontinuation

Investigational Product Product: Ferric maltol oral suspension: oral suspension containing 30 mg elemental iron, in the form of 231.5 mg ferric maltol, in 5 ml suspension.

Ferric maltol oral suspension will be taken every morning and evening at least 30 minutes after a meal. Dosing will be supervised by the parent/legal guardian for children/adolescents throughout the treatment period and recorded on a dosing diary.

Ferric maltol bottles will be labelled for clinical trials use and each bottle will have a unique bottle number which will be utilised in the randomisation procedure.

A final eligibility evaluation must be conducted immediately prior to randomisation.

Reference safety information will be the Investigator Brochure.

Comparator therapy: Ferrous sulfate 125 mg/ml (25 mg/ml elemental iron) oral liquid or equivalent dose will be administered under this protocol. Dosing will be supervised by the parent/legal guardian for children/adolescents throughout the treatment period and recorded on a dosing diary.

Reference safety information will be the currently approved summary of product characteristics.

Statistical methods:

Safety and gastrointestinal tolerability will be compared between ferric maltol oral suspension and ferrous sulfate oral liquid via summaries of treatment emergent adverse events (TEAEs), treatment emergent serious AEs (TESAEs) and treatment-emergent AEs (TEAEs) leading to premature discontinuation of study drug.

Efficacy of ferric maltol will be assessed via the change in Hb concentration from baseline to week 12. If no interim analysis is conducted it will be based on a 95% two-sided confidence interval; If an interim analysis is conducted, a Pocock spending function will be used; the interim analysis will be based on a (100 - 3.45)% two sided confidence interval; if the study does not stop after the interim analysis, the final analysis will be based on a (100 - 2.57)% two sided confidence interval.

For the PK analysis, all analytes in serum will be summarised per PK day, for children and adolescents aged 1 month to 17 years receiving ferric maltol.

In addition, all analytes in urine will be summarised per PK day, for children aged 1 month to less than 2 years.

Full details of the statistical analysis, including the analysis of PK endpoints, will be specified in the statistical analysis plan (SAP).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to comply with the study requirements and to provide written informed consent. In the case of patients under the age of legal consent, the legal guardian(s) must provide informed consent and the patient should provide assent per local and national requirements.
2. Age ≥1 month and ≤17 years at the time of informed consent
3. Subjects must have iron deficiency anaemia defined by the following criteria, as measured by the central laboratory at the screening visit

Haemoglobin thresholds define anaemia by age and gender:

Children (1 m - < 5 yrs) <11.0 g/dl Children (5 yrs - < 12 yrs) <11.5 g/dl Children (12 yrs) <12.0 g/dl Female child (≥13 yrs) <12.0 g/dl Male child (≥13 yrs) <13.0 g/dl and

Ferritin thresholds define anaemia by:

ferritin <30 µg/L, or ferritin <50 µg/L with transferrin saturation (TSAT) <20%, 4. Female subjects of childbearing potential must agree to use a highly effective method of contraception (which includes complete abstinence) until study completion and for at least 4 weeks following their final study visit. Highly effective contraception is defined as a method which results in a low failure rate, i.e., less than 1% per year when used consistently and correctly, such as implants, injectables, some intrauterine contraceptive devices (IUDs), a vasectomised partner and oral contraceptive medications.

The need for contraception and compliance with contraception requirements will be assessed at every visit for adolescent patients, and urine pregnancy testing will be performed at each visit for female subjects of childbearing potential.

Exclusion Criteria:

1. Subject with anaemia due to any cause other than iron deficiency, including, but not limited to,

   a. Untreated or untreatable severe malabsorption syndrome
2. Subjects who have received prior to Screening:

   1. Within 28 days intramuscular or intravenous (IV) injection or administration of depot iron preparation.
   2. Within 7 days single agent iron preparations and during the study.
   3. Within 12 weeks of blood transfusion or is scheduled to have blood transfusion or donation during the study period
   4. Within 28 days erythropoiesis stimulating agents and during the study period
   5. Within 14 days COVID-19 vaccination
3. Subjects with vitamin B12 or folic acid deficiency as determined by the central laboratory screening results. Subjects may start vitamin B12 or folate replacement and rescreen after at least 2 weeks.
4. Has concomitant disease that would significantly compromise iron absorption or absorbed iron utilization such as swallowing disorders and/or extensive small bowel resection.
5. History of active peptic ulcer
6. Has chronic renal disease (eGFR <60 mL/min/m2), as assessed at Screening based on serum creatinine.
7. Known hypersensitivity or allergy to either the active substance or excipients of ferric maltol or ferrous sulfate.
8. Has a known contraindication for treatment with iron preparations, e.g. haemochromatosis, chronic haemolytic disease, sideroblastic anaemia, thalassemia, or lead intoxication induced anaemia.
9. Impaired liver function as indicated by alanine aminotransferase (ALT) or aspartate transaminase (AST)>2.0 times upper normal limit as measured at the Screening visit.
10. Active acute inflammatory disease, including IBD flare or disease exacerbation, which in the opinion of the Investigator, is clinically significant.
11. Active chronic or acute infectious diseases requiring antibiotic treatment.
12. Pregnant or breast feeding.
13. Concomitant medical conditions with extensive active bleeding, other than menstrual cycles; subjects who suffer from menorrhagia may be included at the Investigator's discretion.
14. Scheduled or expected hospitalisation and/or surgery during the course of the study
15. Participation in any other interventional clinical study within 28 days prior to Screening.
16. Diagnosed to be COVID-19 positive by (SARS-CoV-2-RT-PCR positive) within 28 days prior to screening.
17. Cardiovascular, liver, renal, hematologic, psychiatric, neurologic, gastrointestinal, immunologic, endocrine, metabolic, respiratory or central nervous system disease that, in the opinion of the Investigator, may adversely affect the safety of the subject and/or objectives of the study drug or severely limit the lifespan of the subject.
18. Any other unspecified reason that, in the opinion of the Investigator or the Sponsor make the subject unsuitable for enrolment.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-06-09 (Actual); Study Completion 2024-06-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (14):
  - The Center for Clinical Trials, Saraland, Alabama
  - Homestead Research Institute, Homestead, Florida
  - Kissimmee Clinical Research Corp, Kissimmee, Florida
  - Miami Clinical Research, Miami, Florida
  - Medical Research of Westcheste, Miami, Florida
  - Eminent Clinical Research and Associates, North Lauderdale, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - Sierra Clinical Research, Las Vegas, Nevada
  - Levine Cancer Institute, Charlotte, North Carolina
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - BRCR Global Texas, Edinburg, Texas
  - Zion Research, Katy, Texas
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
- BRCR Global Puerto, San Juan, Puerto Rico
- United Kingdom (8):
  - Noah's Ark Children's Hospital for Wales, Cardiff
  - Royal Hospital for Sick Children - Edinburgh, Edinburgh
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - King's College Hospital, London
  - Newham University Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Nottingham University Hospitals, Nottingham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study with a total of 23 clinical sites located in the United States(including Puerto Rico) and United Kingdom. A total of 65 patients were enrolled in the study.
Pre-assignment Details: All eligible subjects aged 1 month to less than 2 years entered a Pre-assignment phase, 1-day Pharmacokinetic assessment day following a single dose of ferric maltol oral suspension.
Groups:
- Ferric Maltol Assigned: 12 weeks open-label Treatment Period for ferric maltol children aged 1 month to <2 years
- Ferric Maltol Randomized: Subjects aged 2-17 will be randomised 1:1 to receive ferric maltol oral suspension or ferrous sulfate oral liquid.
  The first 12 subjects randomised to ferric maltol in each age sub-group (2 - 9 yrs, 10 - 17 yrs respectively) will enter a PK phase with 2 PK days.
  Following PK Day 2 subjects will continue until Week 12. Once the 18 subjects in each age subgroup have finished their PK visits, they will continue until week 12.
  Ferrous sulfate 125 mg/ml (25 mg elemental iron) or equivalent dose was used for all children/adolescents. To maximise the iron replenishment for subjects within this group as well; aged 2
  - 17 yrs were dosed 6 mg/kg to the maximum of 4 ml BID.
- Ferrous Sulfate Randomized: Patients aged 2 to 17 years were randomized 1:1 to receive ferric maltol oral suspension or ferrous sulfate oral liquid.
Period: Overall Study
Arm/Group | Ferric Maltol Assigned | Ferric Maltol Randomized | Ferrous Sulfate Randomized
Started | 4 | 31 | 30
Completed | 3 | 28 | 25
Not Completed | 1 | 3 | 5
Not completed — Withdrawal by Subject | 1 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Maltol Assigned | Ferric Maltol Randomized | Ferrous Sulfate Randomized | Total
Number analyzed (Participants) | 4 | 31 | 30 | 65
Age, Customized [Count of Participants; unit: Participants]
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 4 | 0 | 0 | 4
  Children (2-11 years) | 0 | 10 | 11 | 21
  Adolescents (12-17 years) | 0 | 21 | 19 | 40
  Adults (18-64 years) | 0 | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 23 | 22 | 48
  Male | 1 | 8 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 13 | 12 | 27
  Not Hispanic or Latino | 1 | 18 | 18 | 37
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 9 | 11 | 20
  White | 1 | 18 | 16 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin Concentration
Description: The change in Hb concentration from baseline to Week 12 is summarized based on the mITT Population for each treatment group using descriptive statistics summarized by mean, standard deviation, median, and range (minimum and maximum).
  The Randomized/ITT Population is defined as all patients who were randomized/assigned to treatment arms. The mITT Population is defined as all patients in the ITT Population who received at least 1 treatment dose.
Time Frame: From baseline to week 12.
Population: All patients that finalized Day 84 measurement were reported and analyzed. All patients with a missing Day 84 measurement were imputed using a last observation carried forward approach in which the last available post-baseline measurement was used. Post-baseline measurement was missing in 5 patients in the 2. group (mITT Ferric Maltol) , and 6 patients in the 3. group (mITT Ferrous Sulfate).
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- mITT Ferric Maltol Assigned: The dose of ferric maltol oral suspension that was administered for children aged 1 month to < 2 yrs.
- mITT Ferric Maltol: The dose of ferric maltol oral suspension administered for children aged 2 to - 17 yrs.
- mITT Ferrous Sulfate: Ferrous sulfate oral liquid used for all children/adolescents.
Arm/Group | mITT Ferric Maltol Assigned | mITT Ferric Maltol | mITT Ferrous Sulfate
Number analyzed (Participants) | 3 | 26 | 24
g/L | 17.7 (13.61) | 12.5 (13.89) | 11.5 (13.97)

2. Secondary Outcome: Changes in Ferritin Concentration
Description: Changes in ferritin concentration from baseline to week 12 summarised based on the mITT Population for each treatment group.
  The Randomized/ITT Population is defined as all patients who were randomized/assigned to treatment arms. The mITT Population is defined as all patients in the ITT Population who received at least 1 treatment dose.
Time Frame: From baseline to week 12.
Population: All patients that finalized Day 84 measurement were reported and analyzed. All patients with a missing Day 84 measurement were imputed using a last observation carried forward approach in which the last available post-baseline measurement was used. Post-baseline measurement was missing in 2 patients in the 3. group (mITT Ferrous Sulfate).
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | mITT Ferric Maltol Assigned | mITT Ferric Maltol | mITT Ferrous Sulfate
Number analyzed (Participants) | 3 | 31 | 28
μg/L | 6.3 (8.74) | 8.1 (11.06) | 20.6 (30.97)

3. Secondary Outcome: Change in Iron Concentration
Description: Change in iron concentration from baseline to week 12 summarized based on the mITT Population for each treatment group.
  The Randomized/ITT Population is defined as all patients who were randomized/assigned to treatment arms. The mITT Population is defined as all patients in the ITT Population who received at least 1 treatment dose.
Time Frame: From baseline to week 12.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | mITT Ferric Maltol Assigned | mITT Ferric Maltol | mITT Ferrous Sulfate
Number analyzed (Participants) | 3 | 31 | 28
μmol/L | 1.07 (0.577) | 5.77 (8.518) | 3.64 (8.911)

4. Secondary Outcome: Change in the Percentage of Transferrin Saturation
Description: Change from baseline to Day 84 summarized based on the mITT Population for each treatment group.
  The Randomized/ITT Population is defined as all patients who were randomized/assigned to treatment arms. The mITT Population is defined as all patients in the ITT Population who received at least 1 treatment dose.
Time Frame: From baseline to week 12.
Population: All patients that finalized Day 84 measurement were reported and analyzed. All patients with a missing Day 84 measurement were imputed using a last observation carried forward approach in which the last available post-baseline measurement was used. Post-baseline measurement was missing in 1 patient in the 1. group (mITT Ferric Maltol Assigned) and 2 patients in the 3. group (mITT Ferrous Sulfate).
Measure: Mean (Standard Deviation); unit: Percentage of Transferrin Saturation
Arm/Group | mITT Ferric Maltol Assigned | mITT Ferric Maltol | mITT Ferrous Sulfate
Number analyzed (Participants) | 2 | 31 | 28
Percentage of Transferrin Saturation | 2.0 (0.00) | 7.7 (10.14) | 6.5 (12.39)

5. Secondary Outcome: Cmax for Plasma Maltol Glucuronide
Description: Measured maximum plasma concentration (Cmax) (ng/mL) for plasma maltol glucuronide after a single dose of ferric maltol oral suspension on Visit 2 (PK Day 1) and after twice daily administrations for at least 6 days, on Visit 3 (PK Day 2) after a single morning dose.
  Because of the limitations of PK sampling in the pediatric patient population, data from multiple patients in the same treatment and age group had to be combined, using the naïve pooled approach, to achieve a complete set of observations over time for PK analysis. The data did not support PK parameters generation using noncompartmental analysis (NCA) without combining patients. Using validated PK software WinNonlin, the 'sparse sampling' option was utilized to treat the data as one virtual subject and thus the resulting data did not support reliable error estimates of the PK parameters.
Time Frame: PK parameters assessed at Day 1 (Visit 2) and Day 7-10 (Visit 3).
Population: A total of 20 patients in the ferric maltol group were included in the PK Population. Of these patients, there were 7 patients (3 female patients and 4 male patients) who were 2 to 9 years of age, 3 patients (all female patients) who were 10 to 17 years of age and who received 15 mg BID of ferric maltol, and 10 patients (9 female patients and 1 male patient) who were 10 to 17 years of age and who received 30 mg BID of ferric maltol.
Measure: Number; unit: ng/mL
Groups:
- PK Population Ferric Maltol 15mg (2-9 y) Day 1; PK Population Ferric Maltol 15mg (10-17 y) Day 1; PK Population Ferric Maltol 30mg (10-17 y) Day 1; PK Population Ferric Maltol 15mg (2-9 y) Day 7-10; PK Population Ferric Maltol 15mg (10-17 y) Day 7-10; PK Population Ferric Maltol 30mg (10-17 y) Day 7-10: The PK Population is defined as all randomized/assigned patients who had at least 1 dose of study drug and who had at least 1 evaluable post-dose PK sample.
Arm/Group | PK Population Ferric Maltol 15mg (2-9 y) Day 1 | PK Population Ferric Maltol 15mg (10-17 y) Day 1 | PK Population Ferric Maltol 30mg (10-17 y) Day 1 | PK Population Ferric Maltol 15mg (2-9 y) Day 7-10 | PK Population Ferric Maltol 15mg (10-17 y) Day 7-10 | PK Population Ferric Maltol 30mg (10-17 y) Day 7-10
Number analyzed (Participants) | 7 | 3 | 10 | 7 | 3 | 10
ng/mL | 4350 (NA) | 6810 (NA) | 6420 (NA) | 4250 (NA) | 5940 (NA) | 8160 (NA)

6. Secondary Outcome: Tmax for Plasma Maltol Glucuronide
Description: Time to maximum plasma concentration (Tmax) (h) for plasma maltol glucuronide after a single dose of ferric maltol oral suspension on Visit 2 (PK Day 1) and after twice daily administrations for at least 6 days, on Visit 3 (PK Day 2) after a single morning dose.
  Because of the limitations of PK sampling in the pediatric patient population, data from multiple patients in the same treatment and age group had to be combined, using the naïve pooled approach, to achieve a complete set of observations over time for PK analysis. The data did not support PK parameters generation using noncompartmental analysis (NCA) without combining patients. Using validated PK software WinNonlin, the 'sparse sampling' option was utilized to treat the data as one virtual subject and thus the resulting data did not support reliable error estimates of the PK parameters.
Time Frame: PK parameters assessed at Day 1 (Visit 2) and Day 7-10 (Visit 3).
Population: as for outcome 5
Measure: Number; unit: h
Arm/Group | PK Population Ferric Maltol 15mg (2-9 y) Day 1 | PK Population Ferric Maltol 15mg (10-17 y) Day 1 | PK Population Ferric Maltol 30mg (10-17 y) Day 1 | PK Population Ferric Maltol 15mg (2-9 y) Day 7-10 | PK Population Ferric Maltol 15mg (10-17 y) Day 7-10 | PK Population Ferric Maltol 30mg (10-17 y) Day 7-10
Number analyzed (Participants) | 7 | 3 | 10 | 7 | 3 | 10
h | 1.00 (NA) | 2.13 (NA) | 0.52 (NA) | 0.98 (NA) | 2.78 (NA) | 3.63 (NA)

7. Secondary Outcome: AUC0-t for Plasma Maltol Glucuronide
Description: Area under the plasma concentration-time curve from pre-dose (time 0) to the time of last quantifiable plasma concentration for plasma maltol glucuronide (AUC0-t) (hxng/mL) after a single dose of ferric maltol oral suspension on Visit 2 (PK Day 1) and after twice daily administrations for at least 6 days, on Visit 3 (PK Day 2) after a single morning dose.
  Because of the limitations of PK sampling in the pediatric patient population, data from multiple patients in the same treatment and age group had to be combined, using the naïve pooled approach, to achieve a complete set of observations over time for PK analysis. The data did not support PK parameters generation using noncompartmental analysis (NCA) without combining patients. Using validated PK software WinNonlin, the 'sparse sampling' option was utilized to treat the data as one virtual subject and thus the resulting data did not support reliable error estimates of the PK parameters.
Time Frame: PK parameters assessed at Day 1 (Visit 2) and Day 7-10 (Visit 3).
Population: as for outcome 5
Measure: Number; unit: hxng/mL
Groups:
- PK Population Ferric Maltol 15mg (2-9 y) Day 1 Subject analysis; PK Population Ferric Maltol 15mg (10-17 y) Day 1; PK Population Ferric Maltol 30mg (10-17 y) Day 1; PK Population Ferric Maltol 15mg (2-9 y) Day 7-10; PK Population Ferric Maltol 15mg (10-17 y) Day 7-10; PK Population Ferric Maltol 30mg (10-17 y) Day 7-10: The PK Population is defined as all randomized/assigned patients who had at least 1 dose of study drug and who had at least 1 evaluable post-dose PK sample.
Arm/Group | PK Population Ferric Maltol 15mg (2-9 y) Day 1 Subject analysis | PK Population Ferric Maltol 15mg (10-17 y) Day 1 | PK Population Ferric Maltol 30mg (10-17 y) Day 1 | PK Population Ferric Maltol 15mg (2-9 y) Day 7-10 | PK Population Ferric Maltol 15mg (10-17 y) Day 7-10 | PK Population Ferric Maltol 30mg (10-17 y) Day 7-10
Number analyzed (Participants) | 7 | 3 | 10 | 7 | 3 | 10
hxng/mL | 7670 (NA) | 12000 (NA) | 14600 (NA) | 5900 (NA) | 8070 (NA) | 16700 (NA)

8. Secondary Outcome: Cmax for Baseline Corrected Serum Iron
Description: Measured maximum plasma concentration (Cmax) (μg/dL) for baseline corrected serum iron after a single dose of ferric maltol oral suspension on Visit 2 (PK Day 1) and after twice daily administrations for at least 6 days, on Visit 3 (PK Day 2) after a single morning dose.
  Because of the limitations of PK sampling in the pediatric patient population, data from multiple patients in the same treatment and age group had to be combined, using the naïve pooled approach, to achieve a complete set of observations over time for PK analysis. The data did not support PK parameters generation using noncompartmental analysis (NCA) without combining patients. Using validated PK software WinNonlin, the 'sparse sampling' option was utilized to treat the data as one virtual subject and thus the resulting data did not support reliable error estimates of the PK parameters.
Time Frame: PK parameters assessed at Day 1 (Visit 2) and Day 7-10 (Visit 3).
Population: as for outcome 5
Measure: Number; unit: μg/dL
Arm/Group | PK Population Ferric Maltol 15mg (2-9 y) Day 1 | PK Population Ferric Maltol 15mg (10-17 y) Day 1 | PK Population Ferric Maltol 30mg (10-17 y) Day 1 | PK Population Ferric Maltol 15mg (2-9 y) Day 7-10 | PK Population Ferric Maltol 15mg (10-17 y) Day 7-10 | PK Population Ferric Maltol 30mg (10-17 y) Day 7-10
Number analyzed (Participants) | 7 | 3 | 10 | 7 | 3 | 10
μg/dL | 87.0 (NA) | 40.0 (NA) | 119 (NA) | 96.5 (NA) | 21.0 (NA) | 364 (NA)

9. Secondary Outcome: Tmax for Baseline Corrected Serum Iron
Description: Time to maximum plasma concentration (Tmax) (h) for baseline corrected serum iron after a single dose of ferric maltol oral suspension on Visit 2 (PK Day 1) and after twice daily administrations for at least 6 days, on Visit 3 (PK Day 2) after a single morning dose.
  Because of the limitations of PK sampling in the pediatric patient population, data from multiple patients in the same treatment and age group had to be combined, using the naïve pooled approach, to achieve a complete set of observations over time for PK analysis. The data did not support PK parameters generation using noncompartmental analysis (NCA) without combining patients. Using validated PK software WinNonlin, the 'sparse sampling' option was utilized to treat the data as one virtual subject and thus the resulting data did not support reliable error estimates of the PK parameters.
Time Frame: PK parameters assessed at Day 1 (Visit 2) and Day 7-10 (Visit 3).
Population: as for outcome 5
Measure: Number; unit: h
Groups:
- PK Population Ferric Maltol 30mg (10-17 y) Day 7-10: The PK Population is defined as all randomized/assigned patients who had at least 1 dose of study drug and who had at least 1 evaluable post-dose PK sample (applicable only for the Ferric Maltol group).
  A total of 20 patients in the ferric maltol group were included in the PK Population. Of these patients, there were 7 patients (3 female patients and 4 male patients) who were 2 to 9 years of age, 3 patients (all female patients) who were 10 to 17 years of age and who received 15 mg BID of ferric maltol, and 10 patients (9 female patients and 1 male patient) who were 10 to 17 years of age and who received 30 mg BID of ferric maltol.
Arm/Group | PK Population Ferric Maltol 15mg (2-9 y) Day 1 | PK Population Ferric Maltol 15mg (10-17 y) Day 1 | PK Population Ferric Maltol 30mg (10-17 y) Day 1 | PK Population Ferric Maltol 15mg (2-9 y) Day 7-10 | PK Population Ferric Maltol 15mg (10-17 y) Day 7-10 | PK Population Ferric Maltol 30mg (10-17 y) Day 7-10
Number analyzed (Participants) | 7 | 3 | 10 | 7 | 3 | 10
h | 2.37 (NA) | 2.13 (NA) | 2.00 (NA) | 2.10 (NA) | 2.78 (NA) | 6.63 (NA)

10. Secondary Outcome: AUC0-t for Baseline Corrected Serum Iron
Description: Area under the plasma concentration-time curve from pre-dose (time 0) to the time of last quantifiable plasma concentration for baseline corrected serum iron (AUC0-t) (hxng/mL) after a single dose of ferric maltol oral suspension on Visit 2 (PK Day 1) and after twice daily administrations for at least 6 days, on Visit 3 (PK Day 2) after a single morning dose.
  Because of the limitations of PK sampling in the pediatric patient population, data from multiple patients in the same treatment and age group had to be combined, using the naïve pooled approach, to achieve a complete set of observations over time for PK analysis. The data did not support PK parameters generation using noncompartmental analysis (NCA) without combining patients. Using validated PK software WinNonlin, the 'sparse sampling' option was utilized to treat the data as one virtual subject and thus the resulting data did not support reliable error estimates of the PK parameters.
Time Frame: PK parameters assessed at Day 1 (Visit 2) and Day 7-10 (Visit 3).
Population: as for outcome 5
Measure: Number; unit: hxμg/dL
Arm/Group | PK Population Ferric Maltol 15mg (2-9 y) Day 1 | PK Population Ferric Maltol 15mg (10-17 y) Day 1 | PK Population Ferric Maltol 30mg (10-17 y) Day 1 | PK Population Ferric Maltol 15mg (2-9 y) Day 7-10 | PK Population Ferric Maltol 15mg (10-17 y) Day 7-10 | PK Population Ferric Maltol 30mg (10-17 y) Day 7-10
Number analyzed (Participants) | 7 | 3 | 10 | 7 | 3 | 10
hxμg/dL | 64.4 (NA) | 60.1 (NA) | 374 (NA) | 100 (NA) | 1.93 (NA) | 1180 (NA)

ADVERSE EVENTS:
Time Frame: During the 12-week treatment period and within 2 weeks after receiving the last dose of the study drug.
Arm/Group | Ferric Maltol Assigned | Ferric Maltol Randomized | Ferrous Sulfate Randomized
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 2/3 | 4/31 | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Maltol Assigned (N=3) | Ferric Maltol Randomized (N=31) | Ferrous Sulfate Randomized (N=30)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Maltol Assigned (N=3) | Ferric Maltol Randomized (N=31) | Ferrous Sulfate Randomized (N=30)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study is part of a multicenter trial, and Institution may publish the results of its part of the Study in collaboration with the other investigators, but in complete compliance with this section and with the Confidential Information section. After the multicenter publication or twelve (12) months after completion of the Study, whichever occurs first. Sponsor should be informed at least sixty (60) days prior to the planned date of submission or presentation.

DOCUMENTS (2):
  • Study Protocol (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT05126901/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT05126901/SAP_001.pdf